CLINICAL TRIAL: NCT06965400
Title: Comparison of Automatic and Manual Endotracheal Tube Cuff Pressure Monitoring in Pediatric Intensive Care Patients: A Randomized Controlled Cross-Over Study
Brief Title: Comparison of Automatic and Manual Endotracheal Tube Cuff Pressure Monitoring in Pediatric Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Hasan ağın, Prof.Dr, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024/896
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cuff Pressure; Mechanical Ventilation; Pediatric Intensive Care
Keywords: Cuff pressure; Automatic monitoring; Mechanical ventilation

STUDY DESIGN:
Intervention Model Description: 48 hours total (24 hours each phase, manual vs. automatic)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Cuff Pressure Monitoring (Active Comparator): In this arm, cuff pressure was manually measured and adjusted every 2 hours by nurses using a manometer, to maintain a target pressure between 15 and 25 cmH₂O over a 24-hour period.
  Interventions: Device: Automatic Cuff Pressure Control
- Automatic Cuff Pressure Monitoring (Experimental): In this phase, endotracheal tube cuff pressure was continuously monitored using the IntelliCuff® system (Hamilton Medical, Switzerland), which automatically adjusted the pressure to maintain it within the target range of 15-25 cmH₂O. Nurses intervened only if the system alerted due to a deviation.
  Interventions: Device: Automatic Cuff Pressure Control

INTERVENTIONS:
Device: Automatic Cuff Pressure Control — he IntelliCuff® system (Hamilton Medical, Switzerland) continuously monitored and automatically adjusted cuff pressure to keep it within the target range of 15-25 cmH₂O. Manual intervention was only required upon system alert.
  Other Names: IntelliCuff System

SUMMARY:
This prospective, randomized controlled cross-over study compares automatic (IntelliCuff®) and manual methods of endotracheal tube cuff pressure (CP) monitoring in pediatric intensive care patients. The study evaluates the frequency and duration of cuff pressure deviations outside the recommended range (15-25 cmH₂O) and assesses the impact on nursing workload.

DETAILED DESCRIPTION:
Optimal cuff pressure management in pediatric patients undergoing mechanical ventilation is critical to prevent complications such as aspiration pneumonia or tracheal injuries. This study was designed to compare the effectiveness and safety of continuous automatic cuff pressure monitoring using the IntelliCuff® system versus standard manual cuff pressure monitoring performed by nurses every 2 hours.

Patients aged between 1 month and 18 years requiring invasive mechanical ventilation for at least 48 hours participated in a cross-over study at two tertiary pediatric intensive care units. Each patient underwent two consecutive 24-hour monitoring periods: one with automatic cuff pressure monitoring and another with manual monitoring. Data collected included the frequency and total duration of low (<15 cmH₂O) and high (>25 cmH₂O) pressure episodes, number of manual corrections required, and total nursing intervention time.

This study aims to determine whether automatic monitoring provides better control of cuff pressure, reduces the frequency of cuff-related complications, and decreases nursing workload compared to manual monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 month and 18 years who were intubated with a cuffed endotracheal tube and expected to require invasive mechanical ventilation for at least 48 hours were eligible for inclusion

Exclusion Criteria:

* Patients with tracheostomy, known tracheal pathology, extubated within 48 hours, or those requiring frequent ventilator adjustments due to clinical instability were excluded.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Total Time Spent Under Low Cuff Pressure | 24 hours per intervention phase
  TTotal cumulative time (in hours) during which the endotracheal tube cuff pressure remained below 15 cmH₂O throughout the 24-hour monitoring period in each study phase.
Total Time Spent Under High Cuff Pressure | 24 hours per intervention phase
  Total cumulative time (in hours) during which cuff pressure exceeded 25 cmH₂O in either monitoring method.
Number of Manual Corrections Required Number of Manual Corrections Required Number of Manual Corrections Required Number of Manual Corrections Required Number of Manual Corrections Required | 24 hours per intervention phase
  The number of times the cuff pressure had to be manually corrected due to deviations from the target range during each phase.

SECONDARY OUTCOMES:
Total Nursing Intervention Time | 24 hours per intervention phase
  Total time spent by nurses for cuff pressure monitoring and corrections, including routine checks and manual interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Prof.Dr., Study Chair — Dr. Behcet Uz Children's Hospital
Locations (4):
- Turkey (Türkiye) (4):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Cam Sakura Research and Training Hospital, Istanbul
  - Acibadem University, Acibadem Altunizade Hospital, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topjian AA, Raymond TT, Atkins D, Chan M, Duff JP, Joyner BL Jr, Lasa JJ, Lavonas EJ, Levy A, Mahgoub M, Meckler GD, Roberts KE, Sutton RM, Schexnayder SM; Pediatric Basic and Advanced Life Support Collaborators. Part 4: Pediatric Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S469-S523. doi: 10.1161/CIR.0000000000000901. Epub 2020 Oct 21. No abstract available. PMID 33081526
- [Result] Vottier G, Matrot B, Jones P, Dauger S. A cross-over study of continuous tracheal cuff pressure monitoring in critically-ill children. Intensive Care Med. 2016 Jan;42(1):132-3. doi: 10.1007/s00134-015-4103-8. Epub 2015 Oct 29. No abstract available. PMID 26515515
- [Result] Dauvergne JE, Geffray AL, Asehnoune K, Rozec B, Lakhal K. Automatic regulation of the endotracheal tube cuff pressure with a portable elastomeric device. A randomised controlled study. Anaesth Crit Care Pain Med. 2020 Jun;39(3):435-441. doi: 10.1016/j.accpm.2020.04.007. Epub 2020 May 4. PMID 32376293
- [Result] Zhu G, Wang X, Cao X, Yang C, Wang B, Ang Y, Duan M. The effect of different endotracheal tube cuff pressure monitoring systems on postoperative sore throat in patients undergoing tracheal intubation: a randomized clinical trial. BMC Anesthesiol. 2024 Mar 25;24(1):115. doi: 10.1186/s12871-024-02499-5. PMID 38528475
- [Result] Chenelle CT, Oto J, Sulemanji D, Fisher DF, Kacmarek RM. Evaluation of an automated endotracheal tube cuff controller during simulated mechanical ventilation. Respir Care. 2015 Feb;60(2):183-90. doi: 10.4187/respcare.03387. Epub 2014 Nov 25. PMID 25425705
- [Result] Alzahrani AR, Al Abbasi S, Abahoussin OK, Al Shehri TO, Al-Dorzi HM, Tamim HM, Sadat M, Arabi YM. Prevalence and predictors of out-of-range cuff pressure of endotracheal and tracheostomy tubes: a prospective cohort study in mechanically ventilated patients. BMC Anesthesiol. 2015 Oct 15;15:147. doi: 10.1186/s12871-015-0132-7. PMID 26471790